CLINICAL TRIAL: NCT01051674
Title: A Very High Fiber Diet Versus a Low-carbohydrate Diet for Weight Loss in Obese Individuals With or Without Type 2 Diabetes
Brief Title: A Very High Fiber Diet Versus a Low-carbohydrate Diet for Weight Loss
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Lifestyle Center of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 59217
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity; Type 2 diabetes; Fiber; Dietary fiber; Low-carbohydrate diet; High protein diet
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fiber diet (Experimental)
  Interventions: Other: High fiber vs. low-carbohydrate diets
- Low-carbohydrate diet (Experimental)
  Interventions: Other: High fiber vs. low-carbohydrate diets

INTERVENTIONS:
Other: High fiber vs. low-carbohydrate diets — High fiber diet involves at least 40 grams of dietary fiber or more per day for women and at least 50 grams of dietary fiber per day for men. Low-carbohydrate diet involves less than 120 grams of carbohydrate per day for both men and women.

SUMMARY:
Using a 2x2 complete factorial design, approximately 140 obese men and women who may or may not have type 2 diabetes will be randomized to one of two conditions (70 in each condition): (a) a high fiber diet, or (b) a low-carbohydrate diet. Participants will be instructed to follow their assigned diets for 1 year. Outcome measures of interest will include participants' BMI, waist circumference, blood lipids (total, HDL, and LDL cholesterol, and triglycerides), C-reactive protein, and gastrointestinal peptides. Participants will be recruited from the Loma Linda and San Bernardino city area in southern California.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30.0-42.0 kg/m2
* English-speaking

Exclusion Criteria:

* Pregnancy
* Lactation
* Acute or chronic infection
* Type 1 diabetes
* Participation in another trial
* Active cancers
* Currently using Byetta
* Currently on weight loss medication
* Weight loss of more than 4 lbs. within the last 3 months
* Vegan
* Active eating disorder
* Gastrointestinal problems that may be worsened by a high fiber intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Weight | 1 year

SECONDARY OUTCOMES:
Lipid profiles | 1 year
Gastrointestinal hormones | 1 year
Waist circumference | 1 year
C-reactive protein | 1 year
Blood glucose | 1 year
Serum insulin | 1 year
Hemoglobin A1c | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Serena Tonstad, MD, PhD, MPH, Study Chair — Loma Linda University
Locations (1):
- Loma Linda U Medical Center Diabetes Treatment Center, Loma Linda, California, United States